CLINICAL TRIAL: NCT02778724
Title: France PCI Registry : National Observatory of Interventional Cardiology
Status: Recruiting | Type: Observational
Sponsor: Club Régional des Angioplasticiens de la région Centre (Other)
Collaborators: Agence Régional de Santé du Centre (Unknown); Direction Générale de l'Offre de Soins (Other Government); France PCI Association (Unknown)
Responsible Party: Sponsor
Other Study IDs: France PCI
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Interventional; Cardiology; Angioplasty; Coronary; STEMI; Database
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Rigorous clinical practice assessment is a key factor to improve patient's care and prognosis in interventional cardiology (IC). A multicentric IC observational study (CRAC), fully integrated to usual coronary activity report software, started in Centre Val de Loire (CVL) region in 2014.

CRAC observatory was conduced on five IC CathLab of CVL region. Quality of collected data is regularly evaluated and allowed building an exhaustive, and reliable database. This solution could easily be developed in other French regions.

ELIGIBILITY:
Inclusion Criteria:

* Age =>18 years at enrollment
* Patient who have had a coronary angiogram or angioplasty

Exclusion Criteria:

* Patient who didn't want to participated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients aged over 18 undergoing coronary angiogram or angioplasty
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2014-01; Primary Completion 2030-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Census of interventional cardiology activity | 1 year
  Census, follow-up and monitoring of patients during 1 year, after a coronary angioplasty

SECONDARY OUTCOMES:
Optimization of STEMI patient care time | Less than 24 hours
  Manage STEMI < H24 patients, record and monitor time intervals from first pain to first medical contact in order to achieve and maintain the quality of care

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - Research Cardiology Unit / Les hopitaux de Chartres, Le Coudray, Eure Et Loire
  - Centre Hospitalier Henri Mondor d'Aurillac, Aurillac
  - Centre Hospitalier Jacques Coeur de Bourges, Bourges
  - CHU Caen - Hôpital Côte de Nacre, Caen
  - Hôpital Privé Saint-Martin Caen, Caen
  - CHRU Hôpitaux de Tours - Trousseau, Chambray-lès-Tours
  - CHU Gabriel-Montpied de Clermont-Ferrand, Clermont-Ferrand
  - Clinique Bergouignan, Évreux
  - Hôpital Privé de l'Estuaire, Le Havre
  - Groupe Hospitalier du Havre - Hôpital Jacques Monod, Montivilliers
  - CHR Orléans - Hôpital de la Source, Orléans
  - CHU de Rouen - Hôpital Charles-Nicolle, Rouen
  - Clinique Saint-Hilaire - Rouen, Rouen
  - Pôle Santé Oréliance - Clinique de la Reine Blanche, Saran
  - Clinique Saint-Gatien, Tours